CLINICAL TRIAL: NCT04055389
Title: Preventing de Novo Portal Vein Thrombosis With Antithrombin-III in Patients With Cirrhosis: A Randomized, Double-blinded, Placebo - Controlled Trial (PiVoT-AC Trial)
Brief Title: Preventing de Novo Portal Vein Thrombosis With Antithrombin-III in Patients With Cirrhosis
Acronym: PiVoT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Challenges with recruitment
Sponsor: Jonathan Stine (Other)
Collaborators: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Stine, Assistant Professor Medicine, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00013058
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Portal Vein Thrombosis; Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Antithrombin III

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AT-III treatment (Experimental)
  Interventions: Drug: Antithrombin III
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antithrombin III — Patients with reversal of flow or sluggish flow in the main portal vein (<15 cm/s by Doppler ultrasound exam) will be enrolled and randomized to either weekly infusions of AT-III (half-life ~4 days) at a weight-based dosage according to the following formula:
  [Desired level of AT (100%) - Subject level of AT (%)] * subject weight (kg) 1.4
  or placebo for 24 weeks of therapy.
  Arms: AT-III treatment
Other: Placebo — No study drug
  Arms: Placebo

SUMMARY:
To prevent portal vein thrombosis (PVT) in patients with cirrhosis at risk for PVT by pharmacologic prophylaxis with intravenous antithrombin (AT-III).

DETAILED DESCRIPTION:
PVT is a common complication in patients with cirrhosis, affecting 10% to 25% of patients. PVT is a potentially life-threatening occurrence, complicating transplant candidacy and reducing five-year survival. In addition to the mortality risk posed by PVT, microthrombi within the liver have been linked to decompensation due to the phenomenon of parenchymal extinction. Because of the developing understanding of a baseline hypercoagulable state in many cirrhosis patients, recent studies have demonstrated the benefit of prophylactic anticoagulation with enoxaparin in patients with cirrhosis to prevent PVT. In addition to the benefit in reducing PVT, prophylactic anticoagulation was also found to reduce liver decompensation and improve overall survival.

Risk factors for PVT are well described. The strongest independent risk factor for PVT is portal vein velocity. For each 1 cm/s decrease in portal vein velocity, PVT risk increases 16%. Portal vein velocity <15cm/sec is the best-established cutoff for predicting the development of de novo PVT over the ensuing twelve months.

In addition, patients with cirrhosis and venous thromboembolism (PVT, deep vein thrombosis, pulmonary embolus) have abnormally low levels of AT-III. A recent report by the NPB-06 study group suggest that administering intravenous AT-III at dosage of 1500 units/day for five consecutive days in patients with cirrhosis and AT-III <70% serum level is a safe and effective treatment for PVT with promising short-term partial and complete resolution of PVT. Despite this, the role of AT repletion in preventing PVT remains unknown.

ELIGIBILITY:
Inclusion criteria:

Cirrhosis documented by:

* Liver biopsy OR
* Clinical, imaging, and laboratory findings consistent with cirrhosis AND
* Disease process etiologic for cirrhosis (e.g., chronic viral hepatitis, non-alcoholic steatohepatitis, history of alcohol abuse, cholestatic liver disease)

  * Flow in main portal vein less than 15 cm/sec or reversal of flow as assessed by Doppler ultrasonography
  * Age greater than or equal to 18 and less than or equal to 75 years
  * AT-III <70%
  * Platelet count greater than or equal to 55,000 per uL
  * Laboratories reflective of general health status (normal):
* White blood cell count (4-10.4 K/uL)
* Hemoglobin (11.7-15.0 g/dL) and hematocrit (35-44%)
* Creatinine (0.60-1.00 mg/dL) • Child Pugh Turcotte (CPT) Class A cirrhosis

3.2 Exclusion Criteria

* Allergy to AT-III or one of its ingredients
* CPT Class B or C cirrhosis
* Coagulopathy as indicated by International Normalized Ratio (INR) >= 2.2 or an inherited coagulation disorder
* Active hepatitis C infection expecting to initiate HCV therapy within the next two years
* Established PVT or cavernoma
* Transvenous portosystemic shunt (TIPS) placement
* Previous liver transplantation
* Increased risk of bleeding:

  * Active pathological bleeding including subjects with actively bleeding esophageal varices
  * History of intracranial bleeding
  * Unexplained gastrointestinal bleeding
  * Subjects with large esophageal varices, or varices with endoscopic stigmata of bleeding (e.g., red wale sign)
  * Subjects with gastric or intestinal varices
  * Subjects who are taking medicines that increase the risk of thrombosis (e.g. tamoxifen)
  * Subjects with any clinically significant bleeding within the last one month
  * Need for therapeutic anticoagulation for another indication
  * Concurrent use of antiplatelet medications excluding aspirin 81 mg once daily as aspirin at this dosage does not increase bleeding when given concomitantly with AT-III
* Pregnancy or breastfeeding
* Recent major surgery within six weeks
* Inability or unwilling to give informed consent
* Hepatocellular carcinoma [diagnosed by cross-sectional imaging, e.g., computed tomography (CT) or magnetic resonance imaging (MRI)] or another active malignancy
* Predicted lifespan less than two years
* Severe concurrent disease threatening successful completion of the trial in the opinion of the study principle investigator
* Ongoing substance abuse as judged by the study principal investigator and confirmed by an eight-panel urine drug test at screening
* Significant alcohol consumption (20g/day for women and 30g/day for men)
* Human Immunodeficiency Virus infection
* Worsening liver function based on the two initial laboratory values used to establish baseline laboratory measurements (section 7.2.2 Monitoring and Intervention Plan for Drug-induced Liver Injury)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Development of PVT | up to 72 weeks
  incident of PVT measured by ultrasound at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No